CLINICAL TRIAL: NCT02649140
Title: The Effect of Vinegar Consumption on 24-hour Urinary Risk Factors Associated With Calcium Oxalate Urinary Stone Formation: a Randomised Controlled Trial
Brief Title: Effect of Vinegar Consumption on 24-hour Urinary Risk Factors Associated With Stone Formation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President of the Hospital, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MRER(52)2015
Record Dates: First submitted 2015-12-31; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Urolithiasis
Keywords: 24-hour urine; Calcium oxalate; Vinegar
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (No Intervention): Group1 is control group and participants do not need intervention.
- Group 2 (Experimental): Group 2 is vinegar Group and participants in this group are asked to drink 15ml vinegar(Ninghuafu, Sanxi, China)after dinner at noon and evening respectively for a period of four weeks.
  Interventions: Dietary Supplement: Vinegar group

INTERVENTIONS:
Dietary Supplement: Vinegar group — Each participant in vinegar group drink 15ml vinegar(Ninghuafu,Sanxi,China)after dinner at noon and evening respectively for a period of four weeks.
  Arms: Group 2

SUMMARY:
Purpose:

The aim of this present study is to investigate the effect of vinegar consumption on 24-hour urinary risk factors associated with calcium oxalate urinary stone formation and blood biochemical parameters.

Methods:

The investigators will recruit 50 healthy young student volunteers in this study. By simple random sampling technique, volunteers will be allocated to two groups (group 1, control group; group 2, vinegar group).Each participant in vinegar group drink 15ml vinegar ( Ninghuafu, Sanxi, China) at noon and evening respectively for a period of four weeks.The end point of this study is comparison the outcomes of 24-hour urine and blood biochemical parameters between different group and point-in-time.

DETAILED DESCRIPTION:
Purpose:

The written history of vinegar use in China was more than 5,000 years,and it was used as health care products since ancient times. In addition of the main component of acetic acid, it also contains other acids, esters, polyphenols and other active substances.Previous studies have reported some effects of vinegar, such as delays gastric emptying,relieves fatigue, regulates blood glucose and lipid metabolism, antioxidant, reduces blood pressure and so on. The China national epidemiological study of urolithiasis which was conducted from May 2013 through July 2014 indicated that vinegar may be protective against the formation of urolithiasis (has not been published). Animal experiments showed that vinegar could inhibit oxalate calcium crystal formation in rat kidneys (has not been published). Consequently, we performed this randomized controlled trial to investigate the effect of vinegar consumption on 24-hour urinary risk factors associated with calcium oxalate urinary stone formation and blood biochemical parameters.

Methods:

Study design and participants: We will recruit 50 healthy young student volunteers in this study. The inclusion criteria are male who age 18-35 years, and those with normal renal function,without urolithiasis and congenital urinary tract abnormalities. The exclusion criteria include hematuria, urinary tract infection and have a history of kidney or urinary diversion. We exclude male older than 35 years because usually they have to work and not easy to collect 24-hour sample. The reason of excluding female is that the trail will last four weeks and women's menstrual cycle could affect 24-hour urine collection.

Randomisation:

Trained research clinicians enroll volunteers in a university nearby our hospital. Volunteers will be allocated in a 1:1 ratio to control group(group 1) or vinegar group(group 2) by simple random sampling technique, which is conducted by clinical trial office in urology department of our hospital in Guangzhou, China.

Procedures: Each participant in vinegar group drink 15ml vinegar ( Ninghuafu, Sanxi, China) after dinner at noon and evening respectively for a period of four weeks,and participants in control group do not need intervention.All of participants drink vinegar under the surveillance of research clinicians.

Data collection:

Baseline data will be collected before randomization in our hospital. The baseline data protocol includes urinary ultrasonography, spot urine examines, 24-hour urine analysis and blood chemical examines. The parameters of 24-hour urine analysis include Ph, volume, creatinine, oxalate, citrate, phosphate, uric acid, calcium, magnesium, sodium and chloride. The standard blood analysis protocol included routine haematology, fasting serum glucose, creatinine, urea, uric acid, high-density lipoprotein, low-density lipoprotein, triglycerides, alanine transaminase(ALT), total protein(TP), albumin, glutamyltransferase (GGT) , serum total bile acid, cholesterol, sodium, potassium, calcium and chloride ions. Another tube of blood samples are freeze in -80 degree refrigerator for further analysis of oxidation of blood protein product(AOPP), malondialdehyde(MDA), glutathion peroxidase(GSH-PX), superoxide dismutase(SOD) and catalase activity(CAT).

Follow-up data include 24-hour urine analysis on the 7th, 14th, 21th and 28th day during this period and blood biochemical examines on the 29th day. The protocol of 24-hour urine and blood chemical examines is the same with baseline data. And participants will be asked to make a record of meals for seven days.The ANOVA for repeated measures is used to perform the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Normal renal function.
* Those without urolithiasis
* Those without congenital urinary tract abnormalities.

Exclusion Criteria:

* Those with hematuria
* Those with urinary tract infection
* Those have a history of kidney or urinary diversion.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change of 24-hour urinary risk factors associated with calcium oxalate urinary stone formation | One day before drinking vinegar(the 0th day)and on the 7th,14th,21th and 28th day after drinking vinegar.
  To compare the change of 24-hour urinary risk factors associated with calcium oxalate urinary stone formation which include Ph, volume, creatinine, oxalate, citrate, phosphate, uric acid, calcium, magnesium, sodium and chloride of 24-hour urine between two groups on the 7th,14th,21th and 28th day after drinking vinegar.

SECONDARY OUTCOMES:
Change of blood biochemical parameters | One day before drinking vinegar(the 0th day)and on the 29th day after drinking vinegar.
  To compare the change of blood biochemical parameters which include fasting serum glucose, creatinine, urea, uric acid, high-density lipoprotein, low-density lipoprotein, triglycerides,serum total bile acid, cholesterol, sodium, potassium, calcium and chloride ions before grouping and on the 28th day after drinking vinegar.

OTHER OUTCOMES:
Change of blood oxidative stress markers | One day before drinking vinegar(the 0th day) and on the 29th day after drinking vinegar.
  To compare the change of blood oxidative stress markers which include blood protein product(AOPP),MDA,glutathion peroxidase(GSH-PX),superoxide dismutase(SOD) and catalase activity(CAT) before grouping and on the 28th day after drinking vinegar.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hlebowicz J, Darwiche G, Bjorgell O, Almer LO. Effect of apple cider vinegar on delayed gastric emptying in patients with type 1 diabetes mellitus: a pilot study. BMC Gastroenterol. 2007 Dec 20;7:46. doi: 10.1186/1471-230X-7-46. PMID 18093343
- [Background] Mitrou P, Raptis AE, Lambadiari V, Boutati E, Petsiou E, Spanoudi F, Papakonstantinou E, Maratou E, Economopoulos T, Dimitriadis G, Raptis SA. Vinegar decreases postprandial hyperglycemia in patients with type 1 diabetes. Diabetes Care. 2010 Feb;33(2):e27. doi: 10.2337/dc09-1354. No abstract available. PMID 20103553
- [Background] Setorki M, Asgary S, Eidi A, Rohani AH, Khazaei M. Acute effects of vinegar intake on some biochemical risk factors of atherosclerosis in hypercholesterolemic rabbits. Lipids Health Dis. 2010 Jan 28;9:10. doi: 10.1186/1476-511X-9-10. PMID 20109192
- [Background] Nishidai S, Nakamura Y, Torikai K, Yamamoto M, Ishihara N, Mori H, Ohigashi H. Kurosu, a traditional vinegar produced from unpolished rice, suppresses lipid peroxidation in vitro and in mouse skin. Biosci Biotechnol Biochem. 2000 Sep;64(9):1909-14. doi: 10.1271/bbb.64.1909. PMID 11055395
- [Background] Kondo S, Tayama K, Tsukamoto Y, Ikeda K, Yamori Y. Antihypertensive effects of acetic acid and vinegar on spontaneously hypertensive rats. Biosci Biotechnol Biochem. 2001 Dec;65(12):2690-4. doi: 10.1271/bbb.65.2690. PMID 11826965
- [Background] Johnston CS, Steplewska I, Long CA, Harris LN, Ryals RH. Examination of the antiglycemic properties of vinegar in healthy adults. Ann Nutr Metab. 2010;56(1):74-9. doi: 10.1159/000272133. PMID 20068289
- [Background] Mitrou P, Petsiou E, Papakonstantinou E, Maratou E, Lambadiari V, Dimitriadis P, Spanoudi F, Raptis SA, Dimitriadis G. Vinegar Consumption Increases Insulin-Stimulated Glucose Uptake by the Forearm Muscle in Humans with Type 2 Diabetes. J Diabetes Res. 2015;2015:175204. doi: 10.1155/2015/175204. Epub 2015 May 6. PMID 26064976